CLINICAL TRIAL: NCT01704534
Title: A Prospective Proof of Concept Study to Evaluate the Potential Efficacy of Ustekinumab in Patients With Moderate to Severe Hidradenitis Suppurativa (Acne Ectopica)
Brief Title: A Proof of Concept Study to Evaluate the Effectiveness of Ustekinumab in Hidradenitis Suppurativa
Acronym: HiTS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Janssen-Cilag B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 662507; 2011-002091-16 (EudraCT Number)
Record Dates: First submitted 2012-08-07; First posted 2012-10-11 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis suppurativa; Acne ectopica; Inverse acne; Ustekinumab; Stelara
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ustekinumab (Experimental): Ustekinumab 45 mg or 90 mg (dependent on patient's weight) administered on weeks 0-4-16-28
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — subcutaneous injections of 45 mg or 90 mg (if the participant weighs more than 100 kg) on weeks 0 - 4 - 16 - 28
  Other Names: Stelara

SUMMARY:
The purpose of this study is to determine whether ustekinumab is effective in the treatment of moderate to severe hidradenitis suppurativa.

DETAILED DESCRIPTION:
An open label prospective study is performed to investigate the effectiveness and safety of ustekinumab in hidradenitis suppurativa. Twenty patients will be included. They will receive ustekinumab 45 or 90 mg on weeks 0-4-16-28. Patients will be followed up untill week 40.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Hidradenitis suppurativa Hurley stage II or III
* No response to conventional local and oral antibiotics, or immunnesuppressive medication, or TNF-alpha inhibitors or surgery
* The patient has to be able to complete a dutch questionnaire
* Informed consent must be obtained

Exclusion Criteria:

* Not able to complete a Dutch questionnaire
* Pregnancy or breast feeding
* Active hepatitis B or C infection, HIV or tuberculosis
* Treatment with biologics or other immunosuppressive medicine in the previous 3 months
* Malignancies in the last 10 years with the exception of basal cell carcinoma
* Demyelinating disorders
* Heart failure
* Known allergy to ustekinumab or to its preservatives
* Live vaccins in the next 3 months Sever liver or renal failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-05; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in Sartorius score | 76 weeks
  Clinical response is defined as an improvement of the Sartorius score of at least 50%

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Horváth, MD-PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Netherlands